CLINICAL TRIAL: NCT04307303
Title: A Randomised Sham-controlled, Proof of Principle Study of Abdominal Functional Electrical Stimulation (ABFES) for Bowel Management in Spinal Cord Injury (SCI)
Brief Title: Electrical Stimulation of Abdominal Muscles for Bowel Management in People With Spinal Cord Injury
Acronym: BOWMAN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Salisbury NHS Foundation Trust (Other Government)
Collaborators: Inspire Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BOWMAN
Record Dates: First submitted 2020-03-11; First posted 2020-03-13 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Neurogenic Bowel
MeSH Terms: conditions — Neurogenic Bowel

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Abdominal functional electrical stimulation (Experimental)
  Interventions: Device: abdominal functional electrical stimulation
- Low dose abdominal functional electrical stimulation arm (Sham Comparator)
  Interventions: Device: abdominal functional electrical stimulation

INTERVENTIONS:
Device: abdominal functional electrical stimulation — functional electrical stimulation of the abdominal muscles
  Other Names: ABFES

SUMMARY:
A well-managed bowel program is an essential part of daily life for many people with a SCI. Nevertheless, constipation is frequently reported (42-95%). Constipation embraces a spectrum of harms including both physical & psychological distress. Initial exploratory studies suggest abdominal FES may be useful for decreasing overall bowel management time, decreasing colonic transit time and reducing discomfort. The current study will seek to reproduce previous findings in a 12 week study, using overall bowel management time as a benchmark for establishing proof of principle. The study will include 36 people with a spinal cord injury aged 18 and over with an above T12 injury, a complete or incomplete lesion in a medically stable condition, one year or more after injury. Participants will be randomised into two groups. One group will receive abdominal electrical stimulation and the other group low dose abdominal electrical stimulation. Participants will be asked to keep a bowel diary and complete questionnaires examining quality of life and bowel management.

ELIGIBILITY:
* Inclusion Criteria:
* People with a diagnosis of spinal cord injury
* Age =>18 years of age
* Injury level at or above T12
* complete or incomplete spinal cord lesion
* Medically stable condition
* Reflex bowel
* =>1 year post spinal cord injury
* Exclusion Criteria:
* A history of organic bowel obstruction
* Frequent opioid use,
* Intrathecal baclofen or percutaneous endoscopic gastrostomy
* Inflammatory bowel disease
* Recent abdominal hernia
* Recent gastrointestinal or abdominal surgery
* Lower motor neuron lesions,
* Suspected strictures or fistulae along the gastrointestinal tract
* Physiologic gastrointestinal obstruction.
* Other causes of constipation such as hypothyroidism, hypercalcaemia
* Constipation predominant irritable bowel syndrome prior to diagnosis of SCI
* Involvement in other research trial interventions likely to impact current trial
* Poorly controlled epilepsy,
* Cardiac pacemaker in situ
* Other implanted electrical devices
* Pregnancy or pregnancy planned
* Cancerous tissue in the abdominal region
* Any major skin disorders affecting the abdominal area)
* Severe autonomic dysreflexia (tested at initial assessment).

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2021-07-07 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-06-11 (Actual)

PRIMARY OUTCOMES:
Time required for defecation | 8 weeks
  Time taken to have a bowel movement

SECONDARY OUTCOMES:
Neurogenic bowel dysfunction score | 8 weeks
  Participants can score between 0 and 47 (0=minimum and 47=maximum score) a higher score = greater severity of symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Tamsyn Street, Principal Investigator — Salisbury NHS Foundation Trust
Locations (1):
- Salisbury NHS Foundation Trust, Salisbury, United Kingdom